CLINICAL TRIAL: NCT00691847
Title: Reducing Edema Following Refractive Surgery
Status: Completed | Type: Observational
Sponsor: FORSIGHT Vision3 (Industry)
Responsible Party: Osnat Ehrman, FORSIGHT
Other Study IDs: 0163
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Edema
Keywords: Refractive surgery
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Bilateral post refractive procedure

SUMMARY:
Determine if edema plays a role in refractive surgery

DETAILED DESCRIPTION:
Prospective, comparative study

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent bilateral Refractive surgery for myopic correction.
2. Age 18-60.
3. Evidence of an epithelial defect.
4. Uncorrected visual acuity at study visit better than 20/40
5. Patients able to understand the requirements of the study and willing to follow study instructions, to provide written informed consent to participate, and who agree to comply with all study requirements, including the required study follow-up visits.

Exclusion Criteria:

1. Any other anterior segment abnormality other than that associated with Refractive surgery.
2. Any abnormalities associated with the eye lids.
3. Prior laser treatment of the retina.
4. Any ophthalmic surgery performed within three (3) months prior to study excluding Refractive surgery.
5. Diagnosis of glaucoma.
6. Active diabetic retinopathy.
7. Clinically significant inflammation or infection within six (6) months prior to study.
8. Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator.
9. Participation in any study involving an investigational drug within the past 30 calendar days, or ongoing participation in a study with an investigational device.
10. Intolerance or hypersensitivity to topical anesthetics
11. A medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
12. Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: At least 10 subjects following laser refractive procedure
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Corneal Thickness | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: David Verssano, MD, Principal Investigator — Sorasky Medical Center
Locations (1):
- Sorasky Medical Center, Tel Aviv, Israel